CLINICAL TRIAL: NCT07398482
Title: Feasibility and Preliminary Effectiveness of PrEPwise Intervention on PrEP Initiation Among Black Women in Eastern Virginia
Brief Title: PrEPwise Pilot Among Black Women in Eastern Virginia
Acronym: PrEPwise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-45671; 1K01MH136935-01A1 (NIH)
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections; Sexually Transmitted Infection
Keywords: Pre-Exposure Prophylaxis (PrEP); Community Health Worker (CHW)
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEPwise (PrEPdecision aid) (Experimental): Participants randomized to this arm who are HIV negative will receive the behavioral intervention PrEPwise at the HIV testing clinic.
  Interventions: Behavioral: PrEPwise
- Usual care (Active Comparator): Participants randomized to this arm will receive usual care including standard HIV testing, general HIV information, prep information and information about other available services.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: PrEPwise — PrEPwise intervention is a tablet-based PrEP decision aid delivered by community health workers (CHW) to Black women in the context of their regular HIV testing visits. The intervention includes: Tailored PrEP decision aid providing information on HIV risks, PrEP choices, PrEP costs, how to use PrEP, Adherence guidance, side effects, and access points for obtaining PrEP.
  Arms: PrEPwise (PrEPdecision aid)
Other: Usual care — Usual care includes providing general HIV prevention information, basic PrEP information, and information about other available clinic services.
  Arms: Usual care

SUMMARY:
HIV is a virus that affects many people, but Black women in the U.S. are a population at a much higher risk of getting it compared to white women-about 18 times higher. Pre-exposure prophylaxis (PrEP), a medicine if taken as recommended by a clinician can prevent HIV almost completely (99% effective). The problem is that many Black women, especially those living in the Southern U.S., don't know about this medicine called PrEP or find it hard to access it. To address this, healthcare providers sometimes use "decision aids" which are tools, like brochures or videos, designed to help people understand their medical options and make informed choices based on what's important to them. While these tools have worked well for other health issues, they haven't been widely used for preventing HIV. The challenges are doctors do not have enough time to explain PrEP fully to patients during clinic visits and also some Black women do not trust the healthcare system because of a long history of unfair treatment toward Black communities.

Community health workers (CHWs) are trained health workers from the same communities as their patients and can facilitate their ability to provide culturally appropriate health education and information consistent with patients' values and needs. Because of this, patients are often more comfortable talking to them. This project aims to test the acceptability and effectiveness of a decision tool to be integrated into HIV testing services to help Black women decide if PrEP is right for them. The investigators are calling this intervention PrEPwise. A tool originally designed for women dealing with opioid addiction will be adapted to fit the needs of Black women living in the South. The long-term goal of this project is to make it easier for Black women to learn about PrEP and decide whether to use it, ultimately helping lower the number of new HIV cases in Black women.

DETAILED DESCRIPTION:
The study will follow a type-1 effectiveness-implementation hybrid design as a single-site, single-blinded randomized controlled trial. The following procedures detail the study conduct and masking approach:

Baseline Visit:

* Informed consent process
* Collection of demographic information
* Administration of baseline survey assessing: Perceived HIV risk, PrEP knowledge, PrEP attitudes, PrEP stigma, Discrimination/racism experiences, PrEP norms, Decisional conflict, and Self-efficacy

Randomization and Intervention Delivery:

* Random assignment will be conducted at the individual level with 1:1 allocation using random block sizes of 2
* Randomization assignments will be generated through REDCap's randomization module by the study data analyst
* Only participants will be blinded to their study arm assignment. Study staff delivering the intervention cannot be blinded due to the nature of the behavioral intervention
* Participants will be informed they will receive either enhanced or standard HIV prevention information, without specifying their assigned arm
* The research assistant conducting outcome assessments will be different from the staff delivering the intervention
* Immediate post-intervention survey assessing implementation outcomes

  * Intervention acceptability
  * Intervention feasibility
  * Intervention fidelity 3-Month Follow-up Visit:
* Assessment of effectiveness outcomes:

  * PrEP initiation status
  * PrEP persistence
  * Changes in baseline measures
* Collection of pharmacy fill data. At the 3-month follow-up visit, participants will be asked to self-report whether they initiated PrEP and if they obtained refills.

Additional Procedures:

• Qualitative interviews with a subsample (n=20) of participants to explore perspectives about intervention acceptability, fidelity, barriers, and recommendations for adaptations

The research hypothesis is:

Compared to the control arm, the intervention arm will have (1) a higher percentage of Black women initiate PrEP at 3-months, (2) increased PrEP and HIV risk awareness at 3-month follow-up, (3) reduced HIV PrEP stigma, (4) increased trust in healthcare, and (5) Increased decisional certainty in the choice and intention to use PrEP at 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Black women seeking HIV testing services at the community HIV testing clinic
* Eligible for PrEP according to CDC guidelines
* Willing to be followed for 3 months
* Able to provide contact information
* Able to provide informed consent

Exclusion Criteria:

* Participated in the development of the intervention (provided input in the adaptation of PrEP decision aid)
* Unable to provide informed consent
* Unable to provide contact information
* Currently using PrEP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2027-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Acceptability to Participants of PrEPwise Intervention | 3 months
  Acceptability will be assessed using the client satisfaction survey (CSQ-8), an 8-item instrument with 4 possible responses for each item (1-4). Total scores range from 8 to 32; higher scores indicating greater satisfaction.
Acceptability to Community Health Workers (CHWs) of PrEPwise Intervention | 3 months
  Acceptability will be assessed using the client satisfaction survey (CSQ-8), an 8-item instrument with 4 possible responses for each item (1-4). Total scores range from 8 to 32; higher scores indicating greater satisfaction.
PrEPwise intervention Feasibility | 3 months
  Feasibility will be assessed though process measures including number of participants contacted, number screened for eligibility, number enrolled, and number lost to follow-up.
PrEPwise Intervention Fidelity | 3 months
  Fidelity will be assessed measured using a 10-item fidelity checklist, completed by participants after intervention delivery. Each item on the checklist indicates whether a specific component was delivered as expected (e.g., "The CHW discussed PrEP side effects with me") Items are scores as "yes=1" or "no=0". Total scores range from 0-10, with higher scores indicating higher fidelity to the intervention protocol.

SECONDARY OUTCOMES:
PrEP initiation | 3 months
  PrEP initiation is defined as having at least one PrEP prescription fill during the 3-month period of the study using pharmacy fill data.
PrEP persistence | 3 months
  PrEP persistence is defined as the length of time that a person continued to refill PrEP prescription without an interruption of more than 30 days. PrEP persistence will be assessed using pharmacy refill data obtained at 3-month follow-up. Participants will be categorized as either PrEP-persistence (refilled prescription within 30 days of the previous fill running out) or PrEP non-persistent (gap of >30 days between refills). This binary outcome indicates whether participants maintained continuous PrEP coverage throughout the 3-month study period
Perceived HIV risk | 3 months
  Perceived HIV risk will be measured using the Centers for Disease Control (CDC) 5-item screening tool to determine PrEP eligibility for heterosexual women. Questions assess behavioral risk factors. These questions are: having a sexual partner who is HIV positive, having condomless sex with partners of unknown status, having a bacterial sexually transmitted infection (STI) in the past 6 months, exchanging sex for money or drugs, and injecting drugs. A "yes" response to any of these questions indicates a risk factor. Participants who respond to one or more items are considered at high HIV risk and meet CDC criteria for PrEP eligibility. Higher numbers indicate greater perceived HIV risk.
PrEP knowledge | 3 months
  PrEP knowledge will be assessed using 13-item knowledge scale developed by Walsh et al. (2019). This scale measures knowledge about PrEP through true/false items covering topics including: what PrEP is, how it works, its effectiveness in preventing HIV, who should use, side effects, and how to access it. Items are scored as correct=1 or incorrect/don't know=0. Total scores range from 0 to 13, with higher scores indicating greater knowledge about PrEP.
PrEP attitude | 3 months
  PrEP attitudes will be assessed using 5-item attitudes scale developed by Walsh et al. (2019). This scale measures attitudes toward PrEP use including perceptions of effectiveness, safety, responsibility, adherence burden, and government safety assurance. Responses are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores re calculated by summing item responses, with higher scores indicating more positive attitudes toward PrEP.
PrEP stigma | 3 months
  PrEP stigma will be assessed using 5-item HIV PrEP Stigma scale developed by Walsh et al. (2020). This scale measures perceptions of stigma associated with PrEP use, including judgments about PrEP users, embarrassment about obtaining PrEP, and concerns about disclosure to friends, family, and sexual partners. Responses are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5(strongly agree). Total scores range from 5-25, with higher scores indicating greater perceived PrEP stigma.
Decisional conflict | 3 months
  Decisional conflict will be assessed using the 16-item Decisional Conflict Scale (DCS) developed by O'Connor (1995). The scale measures uncertainty in decision-making across five subscales: uncertainty, feeling uninformed, unclear values, unsupported in decision-making, and ineffective decision-making. Items are rated on a 5-point Likert scale from 1 (strongly agree) to 5 (strongly disagree). Items are summed, divided by 16 then multiplied by 25. Score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Intersectional discrimination experiences | 3 months
  Intersectional discrimination experiences. Intersectional discrimination will be assessed using the validated 31-item Intersectional Discrimination Index (InDI) developed by Scheim and Bauer (2019). The index consists of three subscales measuring: 1) anticipated discrimination (9 items), 2) day-to-day discrimination (9 items), and 3) major discrimination experiences (13 items). Participants rate frequency of discrimination experiences, with higher scores indicting greater experiences of discrimination.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Shangani, PhD, Principal Investigator — Boston University
Locations (1):
- LGBT Life Center (5360 Robin Hood Road, Norfolk, VA 23513, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No